CLINICAL TRIAL: NCT00045097
Title: A Phase II Clinical Trial Of BMS-247550 (NSC 710428), An Epothilone B Analog, In Patients With Breast Carcinoma
Brief Title: Ixabepilone in Treating Patients With Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000256355; NCI-02-C-0229; NCI-5791; NCT00040079 (obsolete NCT alias)
Record Dates: First submitted 2002-09-06; First posted 2003-01-27 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2007-01

CONDITIONS: Breast Cancer
Keywords: male breast cancer; recurrent breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — ixabepilone

INTERVENTIONS:
Drug: ixabepilone

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well ixabepilone works in treating patients with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine any antitumor activity of ixabepilone, in terms of objective response rate, in patients with incurable, locally advanced or metastatic breast cancer.
* Determine the toxicity of this drug in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to prior taxane therapy (yes vs no).

Patients (with or without prior taxane exposure) receive ixabepilone IV over 1 hour on days 1-5. An additional cohort of 37 patients who have received prior taxane therapy are then accrued to receive ixabepilone IV over 1 hour on days 1-3 at a higher starting dose. For all patients, courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity. Patients who receive more than 6 courses with satisfactory response may be treated every 4-5 weeks.

Patients removed for unacceptable toxicty are followed periodically.

PROJECTED ACCRUAL: A total of 105 patients (at least 74 with and 21 without prior taxane exposure) will be accrued for this study within 26 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* adenocarcinoma of the breast

  * Incurable, locally advanced or metastatic disease
  * Primarily stage IV disease, but some inoperable stage III disease may be eligible (e.g., a patient with T4 and/or N2-3 disease who cannot receive doxorubicin or who has already received other therapy) NOTE: *Patients with no available tissue for histologic confirmation but who have documentation of breast surgery and prior chemotherapy are eligible upon approval of the principal investigator
* Measurable disease
* No evidence of CNS metastases by brain MRI or contrast head CT scan

  * CNS metastases controlled by radiotherapy or surgical resection at least 6 months prior to study enrollment are allowed
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female or male

Menopausal status

* Not specified

Performance status

* ECOG 0-2

Life expectancy

* At least 3 months

Hematopoietic

* Granulocyte count at least 1,200/mm^3
* Platelet count at least 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN) (3 times ULN if there is clinical evidence of Gilbert's disease)
* AST and ALT no greater than 2.5 times ULN

Renal

* Creatinine normal OR
* Creatinine clearance greater than 40 mL/min

Other

* No poor medical risk due to other nonmalignant systemic disease
* No active uncontrolled infection
* No sensory, motor, or cranial neuropathy or neuropathic pain grade 2 or greater (unless neuropathy is clearly due to underlying breast cancer)
* No other concurrent serious medical illness
* No prior severe hypersensitivity reactions to agents containing Cremophor EL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior filgrastim (G-CSF), pegfilgrastim, or thrombopoietin (or other platelet growth factors)
* No concurrent immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* No other concurrent chemotherapy for breast cancer

Endocrine therapy

* More than 2 weeks since prior hormonal therapy
* No concurrent hormonal therapy

Radiotherapy

* See Disease Characteristics
* No prior craniospinal radiation
* No prior total body irradiation
* More than 4 weeks since prior radiotherapy

Surgery

* See Disease Characteristics

Other

* No other concurrent investigational drugs
* No concurrent cytochrome p450 3A4 inhibitors, including any of the following:

  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Delaviridine
  * Nelfinavir
  * Amprenavir
  * Ritonavir
  * Indinavir
  * Saquinavir
  * Lopinavir
  * Itraconazole
  * Ketoconazole
  * Fluconazole (> 200 mg/day)
  * Voriconazole
  * Nefazodone
  * Fluvoxamine
  * Verapamil
  * Diltiazem
  * Amiodarone
* Concurrent bisphosphonates for bone metastases allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-05; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Anti-tumor activity as measured by CT scans and bone scans at baseline and every other course
Ixabepilone toxicity as measured by lab studies at baseline and after every course

SECONDARY OUTCOMES:
Tumor tubulin polymerization and p53 expression from biopsy specimens and cDNA microarray testing at baseline and prior to course 2.
Neurotoxicity assessment as measured by Semmes-Weinstein monofilament, sharpened Rombrog, one-legged stance, Jebsen Test of hand function, the grooved pef board , and subjective questionnaires at baseline and prior to every other course

CONTACTS AND LOCATIONS:
Overall Officials: Sandra M. Swain, MD, Principal Investigator — National Cancer Institute (NCI)
Locations (4):
- United States (4):
  - Suburban Hospital, Bethesda, Maryland
  - Oncology Care Associates, Bethesda, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland

REFERENCES:
- [Result] Denduluri N, Low JA, Lee JJ, Berman AW, Walshe JM, Vatas U, Chow CK, Steinberg SM, Yang SX, Swain SM. Phase II trial of ixabepilone, an epothilone B analog, in patients with metastatic breast cancer previously untreated with taxanes. J Clin Oncol. 2007 Aug 10;25(23):3421-7. doi: 10.1200/JCO.2006.10.0784. Epub 2007 Jul 2. PMID 17606971
- [Result] Low J, Croarkin E, Parks R, et al.: Assessment of neurotoxicity in patients receiving BMS-247550 for metastatic breast cancer. [Abstract] Breast Cancer Research and Treatment 85.2: A-358, 2004. Also available online. Last accessed April 22, 2004.